CLINICAL TRIAL: NCT01060917
Title: A Single Center, Open Study in Order to Prove Hypo- and Hyperglycaemic Episodes Using a Non-invasive Glucose Measuring Method in Healthy Volunteers and in Type 1 Diabetic Patients
Brief Title: Glucose Clamp Study to Prove Hypo- and Hyperglycemic Episodes Using a Non-invasive Glucose Monitoring Device
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Profil Institut für Stoffwechselforschung GmbH (Industry)
Collaborators: Pendragon Medical AG Switzerland (Unknown)
Responsible Party: Tim Heise, MD, Profil Institut für Stoffwechselforschung GmbH
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06/0097-Study 4
Record Dates: First submitted 2010-02-01; First posted 2010-02-02 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-01

CONDITIONS: Diabetes Mellitus
Keywords: diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Non-invasive CGMS (continuous glucose monitoring system) — A non-invasive continuous glucose monitoring device measure was applied at the wrist and measure skin glucose as an indirect measure of blood glucose every 10 min.
Procedure: Hyperglycemic and hypoglycemic glucose clamp — The automated glucose clamp technique was used to control glucose levels at baseline glycemia for 1h, hyperglycemia (300 mg/dL) for 1.5 h, and euglycemia (100 mg/dL) for another 1.5 h. A continuous somatostatin infusion was initiated after the 2 h run-in period to suppress endogenous insulin secretion. A glucose solution was infused to increase blood glucose towards the hyperglycemic target level. At the end of the hyperglycemic level the somatostatin infusion was stopped and blood glucose was controlled at the euglycemic target level. On a second study day a hypoglycemic clamp took place, where blood glucose after the run-in period of 2 h was lowered by means of intravenous insulin administration over a period of appr. 30 min to a hypoglycemic level of 45 mg/dL, where it was kept constant for appr. 30 min, after which blood glucose was raised to euglycemia (100 mg/dL) again by means of an intravenous glucose infusion and was kept there for 1.5 hours. .
Device: Non-invasive CGMS (GlucoDay) — The minimally-invasive glucose sensor GlucoDay, was used as a control measure

SUMMARY:
Continuous monitoring of the skin tissue glucose concentration on two different study days using glucose sensors that work on the principle of impedance spectroscopy, with systematic alteration of the blood glucose concentration using the glucose clamp technique in healthy subjects and subjects with type 1 diabetes. Simultaneous determination of electrolyte concentrations in the blood by taking frequent blood samples.

DETAILED DESCRIPTION:
A completely non-invasive continuous glucose monitoring device is considered as a major target of glucose sensor development. The aim of this study is to evaluate the performance of a non-invasive glucose sensor (wristwatch) under controlled conditions (glucose clamp) at hyperglycemia (study day 1) and at hypoglycemia (study day 2). Measurements of the non-invasive glucose monitoring device are compared to those obtained from a minimally invasive glucose monitoring device (GlucoDay, microdialysis principle). In addition, changes in blood electrolyte concentrations as well as their impact on the measurements of the non-invasive glucose sensor are evaluated.

ELIGIBILITY:
Inclusion Criteria:

Healthy male and female volunteers:

* Written informed consent
* Aged between 18 and 40 years
* Body mass index between 18 and 28 kg/m²
* Haemoglobin > 13 g%

Male and female patients with type 1 diabetes:

* Known type 1 diabetes, first manifestation 6 months to 15 years before the start of the study
* HbA1c <= 9%
* Written informed consent
* Aged between 18 and 40 years
* Body mass index between 18 and 28 kg/m²
* Haemoglobin > 13 g%

Exclusion Criteria:

* Uncontrolled arterial hypertension (diastolic blood pressure >100 mmHg and/or systolic blood pressure > 180 mmHg)
* For women, pregnancy or breast-feeding or, for sexually active women of child-bearing age, the use of contraceptive methods considered to be safe (oral contraceptives, IUD, implanted or injected contraceptives, diaphragms, or surgical sterilisation of the patient or her partner)
* Deviations in the lab values (excluding HbA1c), as judged by the investigator to be clinically significant, in particular an increase in transaminases to a level that is two and a half times higher than the upper normal value and a creatinine value that is above the normal range
* Severe acute diseases, as judged by the investigator
* Severe chronic disease, as judged by the investigator
* History of macrovascular illnesses such as pAVK, myocardial infarction
* Known microvascular (diabetic) complications (other than diabetic background retinopathy)
* Positive serology for hepatitis B, hepatitis C or HIV
* Blood donation within 3 months prior to the start of the study and intention of donating blood within 3 months after the end of the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2003-01; Primary Completion 2003-03 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
skin tissue glucose concentration | continuously during the glucose clamp

SECONDARY OUTCOMES:
serum and urine electrolyte concentrations (sodium, potassium, chloride, calcium, magnesium, urea, osmolarity, pH, lactate, p(O2), standard bicarbonate, p(CO2), blood glucose concentration | at 5 min intervals between the individual plateau phases, at 10 min intervals during the plateau phases (of the blood glucose concentration)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Heise, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany

REFERENCES:
- [Derived] Caduff A, Lutz HU, Heinemann L, Di Benedetto G, Talary MS, Theander S. Dynamics of blood electrolytes in repeated hyper- and/or hypoglycaemic events in patients with type 1 diabetes. Diabetologia. 2011 Oct;54(10):2678-89. doi: 10.1007/s00125-011-2210-9. Epub 2011 Jun 15. PMID 21674178